CLINICAL TRIAL: NCT05519449
Title: A Phase 1, Open-Label, Multicenter Study of JANX007 in Subjects With Metastatic Castration-Resistant Prostate Cancer
Brief Title: Study of JANX007 in Subjects With Metastatic Castration-Resistant Prostate Cancer (ENGAGER-PSMA-01)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janux Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PSMA-007-001; ENGAGER-PSMA-01 (Other: Janux Therapeutics., Inc)
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer; Metastatic Castration-resistant Prostate Cancer; Castration Resistant Prostatic Cancer
Keywords: Prostate Cancer; Castration-resistant prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Neoplasms, Castration-Resistant | interventions — darolutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation (Experimental): IV dosing during 21- or 28-day cycles. Dosage per cohort will increase to determine the maximum tolerable dose.
  Interventions: Biological: JANX007
- Backfill Expansion (Experimental): IV dosing during 21- or 28-day cycles. Subjects will be dosed at levels previously declared tolerable.
  Interventions: Biological: JANX007
- Monotherapy Expansion Parts A - D (Experimental): IV dosing during 21- or 28-day cycles. Subjects will be dosed at preliminary recommended phase 2 dose (RP2D).
  Interventions: Biological: JANX007
- Combination Expansion (Experimental): IV dosing during 21- or 28-day cycles. Subjects will be dosed at preliminary recommended phase 2 dose
  Interventions: Biological: JANX007; Drug: Darolutamide

INTERVENTIONS:
Biological: JANX007 — JANX007 is dosed via IV in a 21- or 28-day cycle.
Drug: Darolutamide — Darolutamide is dosed via oral tablets
  Arms: Combination Expansion

SUMMARY:
This study is a first-in-human, Phase 1, open-label, multicenter study to assess the safety, tolerability, pharmacokinetic (PK), pharmacodynamic (PD), and the preliminary efficacy of JANX007 in adults with metastatic castration-resistant prostate cancer (mCRPC).

ELIGIBILITY:
Inclusion Criteria:

* Male ≥18 years of age at the time of signing informed consent
* Histologically or cytologically confirmed adenocarcinoma of the prostate
* For Dose Escalation and Backfill: Having mCRPC that progressed after at least one novel anti-androgen therapy and at least one taxane containing regimen. Participants who have actively refused a taxane containing regimen or are medically unsuitable to receive taxane are eligible
* Adequate organ function
* For Monotherapy Expansion Part a: Have received ≤ 2 anti-androgen therapies in either the HSPC or CRPC setting and no more than 1 prior taxane regimen in the HSPC or CRPC setting. Participants who have actively refused a taxane regimen or are medically unsuitable to receive taxane are eligible.
* For Monotherapy Expansion Part b: Have received ≤ 2 anti-androgen therapies in either the HSPC or CRPC settings
* For Monotherapy Expansion Part d: Have received ≤ 1 anti-androgen therapy and a poly(ADP-ribose) polymerase (PARP) inhibitor for mCRPC and have progressed following treatment with the PARP inhibitor
* For Combination Expansion: Have received ≤ 1 anti-androgen therapy other than darolutamide in the HSPC setting and ≤ 1 taxane in the mCRPC setting. Participants who have actively refused a taxane regimen or are medically unsuitable to receive taxane are eligible.

Exclusion Criteria:

* Prior solid organ transplant
* Prior treatment with PSMA-targeted CAR-T cell therapy or PSMA-CD3, PSMA-CD28 or other CD3 T-cell engaging bispecific antibodies or radioligand therapy
* Clinically significant cardiovascular disease
* For Monotherapy Expansion Part a: Prior receipt of any treatment other than an ARPI or taxane in the mCRPC setting
* For Monotherapy Expansion Part b: Prior receipt of any treatment other than an anti-androgen therapy or prior receipt of a taxane containing regimen or more than 1 prior line of therapy for mCRPC
* For Monotherapy Part d: More than 1 prior line of therapy for mCRPC or prior receipt of any treatment other than an anti-androgen therapy and PARP inhibitor for mCRPC or prior receipt of a taxane in the mCRPC setting
* For Combination expansion: More than 1 prior line of therapy for mCRPC or prior receipt of any treatment other than a taxane for mCRPC or prior receipt of Darolutamide or prior receipt of a taxane for HSPC
* Active clinically significant infection (bacterial, viral, fungal, mycobacteria or other)
* Any medical condition or clinical laboratory abnormality likely to interfere with assessment of safety or efficacy of study treatment

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender Identity
Enrollment: 272 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLT) | 3 years
Incidence of Adverse Events (AE) and Serious Adverse Events (SAE) | 3 years

SECONDARY OUTCOMES:
Area under the concentration time curve to infinity of JANX007 (AUC0-inf) | Pre-dose and at multiple timepoints post-dose on Days 1, 2, 4, 8, 9, 15, 16, 18 up to end of treatment (Up to 3 years)
Maximum observed concentration of JANX007 (Cmax) | Pre-dose and at multiple timepoints post-dose on Days 1, 2, 4, 8, 9, 15, 16, 18 up to end of treatment (Up to 3 years)
Number of participants who develop anti-drug antibodies against JANX007 | Up to 3 years
Duration of Response | Up to 3 years
  Time from documentation of complete response or partial response to disease progression using RECIST v1.1 and PCWG3
Prostate Specific Antigen (PSA) response | Up to 3 years
  Best reduction in PSA level achieved confirmed by a second PSA test ≥21 days later
Radiographic Progression Free Survival (rPFS) | Up to 3 years
  Time from treatment initiation to radiographic evidence of disease progression using RECIST v1.1 and PCWG3
Overall Response Rate | Up to 3 years
  Proportion of participants who achieve a complete response or partial response using RECIST v1.1 and PCWG3
Overall Survival | Up to 3 years
  Time from treatment initiation until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Janux Therapeutics, MD, Study Director — Janux Therapeutics
Locations (35):
- United States (32):
  - University of Alabama at Birmingham Hospital, Birmingham, Alabama
  - Mayo Clinic, Phoenix, Arizona
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA Department of Medicine, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Mayo Clinic, Jacksonville, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Northwell Health R.J. Zuckerberg Cancer Hospital, Lake Success, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University Honickman Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Sarah Cannon Research, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Chris O'Brien Lifehouse (COBLH), Camperdown, New South Wales
  - Southern Oncology Clinical Research Unit (SoCRU), Bedford Park, South Australia
  - Linear Clinical Research Ltd., Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No